CLINICAL TRIAL: NCT06407557
Title: Optimizing Older Adults' Home Space: Feasibility Trial to Reduce Sedentary Behaviour and Increase Physical Activity.
Brief Title: Optimizing Older Adults' Home Space for Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swansea University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2 2023 6667 6123
Record Dates: First submitted 2024-02-08; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Accelerometer (Active Comparator)
  Interventions: Behavioral: Accelerometer
- No arm accelerometer (Active Comparator)
  Interventions: Behavioral: Accelerometer

INTERVENTIONS:
Behavioral: Accelerometer — Use of prompts to enable activity in older adults.

SUMMARY:
There will be a multi-channel approach to recruitment. Currently, ongoing projects within diverse communities lead in Swansea, Bridgend, and Neath Port Talbot will be approached, and this research will recruit alongside these projects. Regional coordinators and sub-coordinators will be contacted for recruitment, to best ensure participating older adults reflect the typical socio-demographics of Wales. This network will help the researchers to reach older adults who previously took part in different projects. Recruitment letter posters/leaflets will be used as an enrolment technique. Furthermore, the researchers will place advertisements across the University using the intranet and work alongside the City and County of Swansea, Neath Port Talbot, and Bridgend Borough Council to recruit using their sport, play, and community networks. The first stage of recruitment involves approaching diverse community organizations to formally request approval to recruit via their contacts. In-stage gatekeepers will be approached by the researcher to seek permission to contact potential participants via their organization. All interested participants will be asked to contact the researcher directly to further discuss the study and indicate their interest. All participants will provide written informed consent to participate in the study before the baseline assessment is conducted. Moreover, each older adult will receive a sleeping log (to record not wearing time), an accelerometer device, and instructions on how to attach and wear the device for 7 consecutive days. The primary researcher will be contacted if older adults have any queries or issues with the device. The participants will be subsequently randomized to an intervention group or comparison group on the basis of 1:1 allocation. All assessments including questionnaires and a 7-day accelerometer assessment will be repeated post-intervention. An Independent t-test will be run to assess the pre-post difference in the effectiveness of the trial in the intervention and comparison groups. The regression model will be applied to assess the impact of covariates with the dependent variables (MVPA, daily step count, self-efficacy, well-being, and sedentary behaviour). Qualitative data analysis of interview data will use reflexive thematic analysis to illustrate common themes regarding the acceptability of the feasibility trial.

DETAILED DESCRIPTION:
There will be a multi-channel approach to recruitment. Currently, ongoing projects within diverse communities lead in Swansea, Bridgend, and Neath Port Talbot will be approached, and this research will recruit alongside these projects. Regional coordinators and sub-coordinators will be contacted for recruitment, to best ensure participating older adults reflect the typical socio-demographics of Wales. This network will help the researchers to reach older adults who previously took part in different projects. Recruitment letter posters/leaflets will be used as an enrolment technique. Furthermore, the researchers will place advertisements across the University using the intranet and work alongside the City and County of Swansea, Neath Port Talbot, and Bridgend Borough Council to recruit using their sport, play, and community networks. Step 1: In step 1 of recruitment, the lead researcher will request approval from the project leads to make a visit to pitch for participants to both explain the study and provide important information to older adults. Interested older adults will be asked to write down their name and preferred contact details in the space provided on the study letters, and to return them to their respective area project lead. Step 2: The researcher will contact interested older adults via email or phone. Older adults who agree to take part will receive participant information sheets, which will be arranged for the researcher to meet them in their home. Step 3: The lead researcher will explain the study process and procedures and answer any questions ensuring the person is fully informed of the nature of the study and how taking part will affect them. Providing the older adult is happy to proceed, they will be given a consent form to sign where the baseline assessment can be undertaken. The first stage of recruitment involves approaching diverse community organizations to formally request approval to recruit via their contacts. Based on the premise that approval is obtained, in-stage gatekeepers will be approached by the researcher to seek permission to contact potential participants via their organization. Gatekeepers will, in no instance, be asked to discuss the study with potential participants. Rather, they will be approached to identify individuals to gain approval to contact individuals to describe the study and share pertinent information. All interested participants will be asked to contact the researcher directly to further discuss the study and indicate their interest. The researcher will organize a time for formal enrolment and induction into the study with the interested older adults. All participants will provide written informed consent to participate in the study before the baseline assessment is conducted. Moreover, each older adult will receive a sleeping log (to record not wearing time), an accelerometer device, and instructions on how to attach and wear the device for 7 consecutive days. The primary researcher will be contacted if older adults have any queries or issues with the device. The participants will be subsequently randomized to an intervention group or comparison group on the basis of 1:1 allocation. All assessments including questionnaires and a 7-day accelerometer assessment will be repeated post-intervention. The normality of the outcome variable will be assessed through a histogram. An Independent t-test will be run to assess the pre-post difference in the effectiveness of the trial in the intervention and comparison groups. The regression model will be applied to assess the impact of covariates with the dependent variables (MVPA, daily step count, self-efficacy, well-being, and sedentary behaviour). Qualitative data analysis of interview data will use reflexive thematic analysis to illustrate common themes regarding the acceptability of the feasibility trial. Using this approach, notes and initial impressions will be taken by the researcher during the interviews. These themes will be tracked and continually revised throughout transcription and later themes are developed based on underlying meaning.

ELIGIBILITY:
Inclusion Criteria:

* All participants aged ≥ 65 years old and able to do their daily living activities.

  * Be able to communicate in English.
  * Self-reported daily sitting time of 6 hours/day

Exclusion Criteria:

* • are not able to cooperate with the research team for the full duration of the project.

  * any exercise contraindications
  * cognitive impairment, or other mental health diagnosis and/or psychological impairment.
  * living in a supported nursing home or in long-term care.
  * participating in daily moderate to vigorous physical activity level (> 150 minutes/week) These criteria were put in place to ensure a group of sedentary older adults who could safely alter their sitting habits in an unsupervised intervention.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 23 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-04-22 (Actual); Study Completion 2024-04-22 (Actual)

PRIMARY OUTCOMES:
Feasibility assessment | 2 months
  Retention = Older adults completed post intervention assessment (semi-structured interviews)/ older adults enrolled * 100

SECONDARY OUTCOMES:
Activity | 2 months
  Activity will be measured with a wrist-worn accelerometer (Actigraph wGT9X Link+, Pensacola, FL).
Self-efficacy | 2 months
  Self-efficacy for activity will be measured using the Self-Efficacy for Exercise Scale. The Self-Efficacy for Exercise Scale is a self-report measure with 5 items assessing one's degree of confidence in the ability to perform activity. The score is the sum of the item responses; higher scores indicate greater self-efficacy.
Sitting Behaviours | 2 months
  Self-Report Habit Index will be used to measure habits associated to SB (Sedentary Behaviour) and PA (Physical Activity), previously validated in studies.
Well-being | 2 months
  The Warwick-Edinburgh Mental Wellbeing Scale, a 14-item self-report measure, will be used to assess well-being. Respondents rate their experience regarding each statement over the last 2 weeks. Each item is scored using a 5-point Likert scale ranging from 1 (none of the time) to 5 (all of the time), with the total score ranging from 14 (low well-being) to 70.
Acceptability | 3 months
  Semi-structured interviews
Uptake | 4 months
  The intervention uptake will be assessed as:
  Uptake = Older adults enrolled/older adults invited to take part in the study * 100
Data Completeness | 3 months
  Data completeness: The data completeness will be assessed as:
  Data completeness = Older adults return to complete accelerometer derived and self-report data/older adults enrolled * 100

CONTACTS AND LOCATIONS:
Locations (1):
- Swansea University, Swansea, United Kingdom

REFERENCES:
- [Derived] Meghani NAA, Hudson J, Stratton G, Mullins J, Sahoo D. A multi-method feasibility trial of a multi-component behaviour change intervention to reduce sedentary behaviour and increase physical activity among ethnically diverse older adults. BMJ Open. 2024 Nov 7;14(11):e084645. doi: 10.1136/bmjopen-2024-084645. PMID 39510783